CLINICAL TRIAL: NCT07395648
Title: Effect of Smartwatch Along With Foundation Model for the Monitoring and Management of Acute Myocardial Infarction Patients During Outpatient Cardiac Rehabilitation After Percutaneous Coronary Intervention: Protocol for a Randomised Controlled Multicentre Trial
Brief Title: Foundation Model for Post-MI Cardiovascular Event Alert Using Huawei Watch
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Collaborators: Beijing Anzhen Hospital Affiliated to Capital Medical University (Unknown); Fengtai Rehabilitation Hospital of Beijing Municipality (Tieying Hospital) (Unknown); Beijing Aerospace General Hospital (Other); First Affiliated Hospital of Harbin Medical University (Other); The Third People's Hospital of Chengdu (Other); Second Hospital of Jilin University (Other); Qilu Hospital of Shandong University (Other); Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Zhang Cuntai, Professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2025S128
Record Dates: First submitted 2026-01-22; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Coronary Artery Disease; Myocardial Infarction
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention I group (the smartwatch with AI assisted group) (Experimental): Subjects in the intervention group will be required to wear a smartwatch continuously for 3 months. For patients in Intervention group, the smartwatch will record the daily activities and sleep status. Furthermore, for patients in Intervention I group, the pre-trained foundation model will generate preliminary diagnostic suggestion based on the data collected by the smartwatch to remind the appearance of heart failure, myocardial ischemia, arrhythmia, abnormal blood pressure, and abnormal cerebral blood supply.
  Interventions: Device: Smartwatch + AI assisted
- Intervention II group (smartwatch assisted group) (Experimental): Subjects in the intervention group will be required to wear a smartwatch continuously for 3 months. For patients in Intervention group, the smartwatch will record the daily activities and sleep status.
  Interventions: Device: Smartwatch only
- Control group ( conventional care) (Active Comparator): Participants will receive routine outpatient CR and follow-up.
  Interventions: Device: Conventional care

INTERVENTIONS:
Device: Smartwatch + AI assisted — All patients will receive routine outpatient CR and follow-up. Subjects in the intervention group will be required to wear a smartwatch continuously for 3 months. For patients in Intervention group, the smartwatch will record the daily activities and sleep status. Furthermore, for patients in Intervention I group, the pre-trained foundation model will generate preliminary diagnostic suggestion based on the data collected by the smartwatch to remind the appearance of heart failure, myocardial ischemia, arrhythmia, abnormal blood pressure, and abnormal cerebral blood supply.
  Arms: Intervention I group (the smartwatch with AI assisted group)
Device: Smartwatch only — All patients will receive routine outpatient CR and follow-up. Subjects in the intervention group will be required to wear a smartwatch continuously for 3 months. For patients in Intervention group, the smartwatch will record the daily activities and sleep status.
  Arms: Intervention II group (smartwatch assisted group)
Device: Conventional care — All patients will receive routine outpatient CR and follow-up.
  Arms: Control group ( conventional care)

SUMMARY:
The goal of this randomized controlled trial is to evaluate whether a HUAWEI smartwatch integrated with a foundation model can enhance daily monitoring and management of AMI patients during outpatient cardiac rehabilitation after PCI.

Can a HUAWEI smartwatch with a foundation model improve daily monitoring/management of post-PCI AMI patients during 3-month outpatient CR, vs routine management or smartwatch without AI? Does the AI-enabled smartwatch (Intervention I) reduce 3-month cardiovascular-related hospital/emergency visits vs the other two groups? Do smartwatches (with/without AI) enhance quality of life and activity function post 3-month CR? Does the AI-enabled smartwatch lower 1-year major adverse cardiovascular events (MACEs) and related hospital/emergency visits vs other groups? How accurate is the AI-enabled smartwatch's alert system (vs hospital diagnostic results) for cardiovascular abnormalities? What is the usability of the AI-enabled smartwatch for patients and doctors?

Participants will:

Sign informed consent; complete baseline exams (MET, SF-36, 6-minute walk, exercise tolerance test) and questionnaires (demographics, medical history, medications).

Receive 3-month outpatient CR. Attend follow-ups; report all adverse events promptly.

Intervention I (AI-Enabled Smartwatch) group Wear the smartwatch continuously for 3 months (sleep wear recommended); actively collect ≥30s ECG via the watch's crown.

Pause activity if heart rate exceeds anaerobic threshold; adjust exercise intensity if METs mismatch prescription.

Contact doctors immediately upon receiving abnormality alerts (e.g., heart failure); follow expert recommendations for further care; complete usability questionnaires.

Intervention II (Non-AI Smartwatch) group Wear the smartwatch continuously for 3 months (sleep wear recommended) to track activity/sleep, monitor real-time heart rate/MET.

Pause activity if heart rate exceeds anaerobic threshold; adjust exercise intensity if METs mismatch prescription.

Control Group Complete routine outpatient CR and follow-ups (no smartwatch use).

ELIGIBILITY:
Inclusion Criteria:

1. Aged more than equal to 18 years, less than 69 years.
2. Discharged within 6 months after PCI for acute myocardial infarction, and haven't received outpatient cardiac rehabilitation;
3. 40%≤EF≤50% and NT-pro BNP ≤500 pg/mL;
4. With the history of hypertension;
5. Voluntarily joined and signed the informed consent.

Exclusion Criteria:

1. With contraindication for rehabilitation activities include: unstable angina, uncontrolled hypertension (systolic blood pressure>180 mmHg and/or diastolic blood pressure>110 mmHg in a quiet state), severe symptomatic heart valve stenosis, uncontrolled heart rate increase (>130 beats/minute), uncontrolled heart failure, third degree atrioventricular block (without pacemaker implantation), active pericarditis or myocarditis, presence of newly formed embolism (pulmonary or systemic circulation), aortic dissection, acute thrombophlebitis, acute systemic disease or fever, other metabolic abnormalities (such as acute thyroiditis, electrolyte imbalance, uncorrected blood glucose abnormalities or insufficient blood volume), and severe psychological disorders;
2. Patients who have a pre-planned staged revascularization procedure (e.g., planned second coronary intervention) following their initial PCI for AMI.
3. Tattoos or other substances that affect optical signals on the wrist.
4. Coronary heart disease patients at high risk.
5. Pregnant women or women planning to become pregnant within the next year.
6. Severe arrhythmia, including third degree atrioventricular block, ventricular escape rhythm, severe sinus bradycardia, sick sinus syndrome, supraventricular tachycardia, ventricular tachycardia, atrial fibrillation, atrial flutter, ventricular fibrillation, ventricular flutter.
7. Physical disability, blindness, and deafness.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1050 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Major adverse events | Three months.
  Occurrence of major adverse events (MI, stroke or death)

SECONDARY OUTCOMES:
Motor function | Three months
  Assessed by metabolic equivalent of task
Quality of life | Three months
  Assessed by 36-Item Short Form Health Survey
Exercise tolerance | Three months
  Assessed by 6-minute walking distance

OTHER OUTCOMES:
Major adverse cardiovascular events-1 year | One year
  The occurrence of major adverse events from baseline to 1 year of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Cuntai Zhang, PhD, Study Chair — Wuhan TongJi Hospital